CLINICAL TRIAL: NCT06563895
Title: A Phase 3, Randomized, Multicenter, Double-Blind, Placebo-Controlled Study of Acoramidis for Transthyretin Amyloidosis Prevention in the Young (ACT-EARLY Trial)
Brief Title: Acoramidis Transthyretin Amyloidosis Prevention Trial in the Young (ACT-EARLY) Study in Asymptomatic Carriers of a Pathogenic TTR Variant
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eidos Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AG10-501; U1111-1307-8107 (Other: WHO); jRCT2071250116 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-08-05; First posted 2024-08-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Amyloidosis; Amyloid Cardiomyopathy; Transthyretin Amyloidosis; Cardiomyopathies; Heart Diseases; Polyneuropathies
Keywords: Amyloidosis; ATTR-CM; ATTR-PN; Transthyretin; Amyloid; TTR
MeSH Terms: conditions — Amyloidosis; Amyloid Neuropathies, Familial; Amyloidosis, Hereditary, Transthyretin-Related; Cardiomyopathies; Heart Diseases; Polyneuropathies; Alzheimer Disease | interventions — attruby

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- acoramidis (Experimental): Participants will receive acoramidis 712 mg orally BID (which is equivalent to 800 mg acoramidis HCl BID)
  Interventions: Drug: Acoramidis
- Placebo (Placebo Comparator): Subjects will receive placebo to match twice daily
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Acoramidis — TTR stabilizer administered orally twice daily (BID)
  Other Names: AG10; ALXN2060
  Arms: acoramidis
Drug: Placebo oral tablet — Non-active control administered orally twice daily (BID)
  Arms: Placebo

SUMMARY:
Transthyretin amyloidosis (ATTR) is a disease where the normally occurring transthyretin (TTR) protein falls apart and forms amyloid, a sticky plaque- like substance that accumulates in different organs in the body and can cause damage to the organ. There are two ways that the TTR protein can fall apart. One way occurs as a person ages, where the normal TTR protein can fall apart and form amyloid that may no longer be sufficiently cleared by the body. This type of ATTR is known as wild-type ATTR (ATTRwt). The other way occurs when a person inherits a defective TTR gene that causes the TTR protein to spontaneously fall apart. This form of the disease is known as variant ATTR (ATTRv) and can be detected in adults by a genetic test of their TTR gene before they age.

Amyloid build-up in the heart causes the heart wall to become thick and stiff and can result in heart failure and even death. Accumulation of TTR amyloid in the heart is known as transthyretin amyloid cardiomyopathy or ATTR-CM. Amyloid can also deposit in the nerve tissues leading to nerve problems. Accumulation of TTR in the nerves is known as transthyretin amyloid polyneuropathy or ATTR-PN.

Acoramidis is an experimental drug designed to bind tightly to TTR in the blood and stabilize its structure, so it does not form the harmful amyloid plaques that can cause damage to organs.

This study is intended to determine if treatment with acoramidis in participants with ATTRv who have not yet developed any symptoms of disease can prevent or delay the development of ATTR-CM or ATTR-PN disease. If adults with an inherited defective TTR gene are treated early before any of the symptoms of disease have developed, it may be possible to delay the onset or prevent the disease entirely.

DETAILED DESCRIPTION:
The AG10-501 ACT-EARLY study is a randomized, multicenter, double-blind, placebo- controlled study of acoramidis for prevention of ATTR (with specific reference to either its cardiomyopathic or polyneuropathic manifestations). Participants will be stratified at randomization.

The study population will be asymptomatic carriers of a known pathogenic TTR gene variant. A participant must be 18 to 75 inclusive years of age, and the age of the participant must be no more than 10 years younger than the predicted age of disease onset (PADO) based either on family history (pedigree analysis) or, if family history is insufficient, based on a TTR Variant Actuarial table from published literature. For example, if PADO for a given individual is found to be 50 years, the age of the participant must be between 40 and 75 years inclusive.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female ≥ 18 to ≤ 75 years of age inclusive.
* Participants must have an established genotype (hetero- or homozygosity) of a TTR gene variant that is known to be pathogenic (eg, V30M/p.V50M, V122I/p.V142I, T60A/p.T80A, or any other pathogenic TTR variant(s)) confirmed by central laboratory prior to randomization.
* Participant's age is no more than 10 years (≤ 10) younger than the PADO.

Key Exclusion Criteria:

* Evidence of ATTR-CM or ATTR-PN.
* Presence of a TTR variant known to be phenotypically protective (eg, T119M, R104H).
* Current or past treatment with other TTR modifying therapies.
* Contraindication to or inability to undergo Cardiac magnetic resonance testing.
* Major organ dysfunction, including: kidney disease, liver disease, heart disease (including cardiomyopathy), neuropathy
* Other diseases or conditions such has cancer within 3 years, untreated hyperthyroidism or hypothyroidism, type 1 diabetes, active hepatitis B or C, HIV.
* Major surgery within the past 3 months or planned during the next 12 months.
* Known hypersensitivity to acoramidis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Time to development of ATTR (ATTR-CM or ATTR-PN, whichever occurs first; centrally adjudicated) | Since randomization up to approximately 7 years or until the study is declared over
  * ATTR-CM defined by biopsy or imaging-based diagnosis
  * ATTR-PN defined by new signs or symptoms and biopsy-based diagnosis

SECONDARY OUTCOMES:
Time to development of ATTR-CM (centrally adjudicated) | Since randomization up to approximately 7 years or until the study is declared over
  ATTR-CM defined by biopsy or imaging-based diagnosis
Time to development of ATTR-PN (centrally adjudicated) | Since randomization up to approximately 7 years or until the study is declared over
  ATTR-PN defined by new signs or symptoms and biopsy-based diagnosis

CONTACTS AND LOCATIONS:
Locations (90):
- United States (37):
  - University of California, San Diego (UCSD) - Medical Center, La Jolla, California
  - University of California, Los Angeles (UCLA) - David Geffen School of Medicine, Los Angeles, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado Anschutz, Aurora, Colorado
  - Yale University School of Medicine - Section of Cardiology, New Haven, Connecticut
  - MedStar Washington Hospital Center - MedStar Heart and Vascular Institute, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Chicago - Medical Center, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University (BU) School of Medicine, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New York University (NYU) School of Medicine - Langone Medical Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Laurelton Heart Specialists, Rosedale, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - National Neuromuscular Research Institute, Austin, Texas
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
- Australia (2):
  - St Vincent's Hospital Sydney, Darlinghurst
  - Westmead Hospital, Westmead
- UZ Leuven, Leuven, Belgium
- Brazil (4):
  - Fundacao Centro Medico de Campinas, Campinas
  - Instituto do Coracao (InCor) do Hospital das Clinicas da FMUSP, Cerqueira César
  - CAPED - Centro Avancado de Pesquisa, Estudos e Diagnostico, Ribeirão Preto
  - Cardiopulmonar da Bahia S.A. (Hospital Cardio Pulmonar), Salvador
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
- Hvitfeldt Poulsen, Aarhus, Denmark
- France (5):
  - CHU Bordeaux - Hopital Pellegrin, Bordeaux
  - AP-HP Hopital Henri Mondor, Créteil
  - AP-HP Hopital Bicetre, Le Kremlin-Bicêtre
  - CHU Rennes, Rennes
  - CHU de Toulouse - Hopital Rangueil, Toulouse
- Germany (2):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Heidelberg, Heidelberg
- Greece (2):
  - Hippokration General Hospital of Athens, Athens
  - General Hospital of Athens - Alexandra, Athens
- Ireland (2):
  - The Mater Misericordiae University Hospital, Dublin
  - Tallaght University Hospital - The Adelaide and Meath Hospital, Dublin
- Italy (6):
  - Azienda Ospedaliero-Universitaria di Bologna IRCCS Policlinico di S.Orsola, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Toscana Gabriele Monasterio per la Ricerca Medica e di Sanità Pubblica - Ospedale San Cataldo, Pisa
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Rome
- Kumamoto University Hospital, Kumamoto, Japan
- University Malaya Medical Centre (UMMC), Kuala Lumpur, Malaysia
- CHU de Fort de France, Fort-de-France, Martinique
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Portugal (2):
  - Unidade Local de Saude de Santa Maria EPE - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saude de Santo Antonio EPE - Hospital de Santo Antonio, Porto
- Singapore General Hospital, Singapore, Singapore
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
- Spain (5):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Universitario Son Llatzer, Palma de Mallorca
  - Hospital Clinico Universitario de Salamanca, Salamanca
- Norrlands universitetssjukhus (University Hospital of Umea), Umeå, Sweden
- Taiwan (3):
  - Changhua Christian Hospital - Taiwan, Changhua
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (2):
  - St. Bartholomew's Hospital, London
  - University College London Hospitals NHS Foundation Trust, London